CLINICAL TRIAL: NCT03995368
Title: New Applications of Neuroplasticity Biomarkers in Veterans With Traumatic Brain Injury or Schizophrenia
Brief Title: Neuroplasticity in TBI and Schizophrenia
Acronym: NVEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D3171-P
Record Dates: First submitted 2019-06-14; First posted 2019-06-24 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Traumatic Brain Injury
Keywords: Schizophrenia; Traumatic Brain Injury; Neuroplasticity; EEG
MeSH Terms: conditions — Schizophrenia; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: All participants will have the same tasks delivered in the same manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- People with Schizophrenia (Experimental): People who have been diagnosed with schizophrenia and meet the investigators' research criteria for symptoms indicative of schizophrenia within their lifetime.
  Interventions: Other: Electroencephalography
- People with TBI (Experimental): People who have been diagnosed with a mild or moderate traumatic brain injury (TBI) and meet research criteria indicative of TBI within their lifetime.
  Interventions: Other: Electroencephalography
- Healthy Controls (Experimental): People without a history of psychiatric illness or TBI and who do not meet research criteria for a psychiatric illness or TBI.
  Interventions: Other: Electroencephalography

INTERVENTIONS:
Other: Electroencephalography — The investigators will use EEG combined with measures of cognition and clinical interviews to explore connections between these measures and electrical activity in the brain in Veterans with a diagnosis of schizophrenia or TBI, and healthy controls.
  Other Names: EEG

SUMMARY:
This proposal will examine measures of neuroplasticity (the brain's ability to alter its function or structure in response to changes in the environment or novel experiences) in Veterans with schizophrenia or traumatic brain injury (TBI). Both conditions are associated with impaired cognition (for example, attention, memory, learning), which is in turn associated with poor community functioning and integration. However, the two disorders differ in their origins: schizophrenia is a neurodevelopmental disorder appearing usually in late adolescence while TBI is an acquired disorder as the result of an injury to the head. Understanding of the root causes of complex cognitive impairments associated with these disorders remains limited. Neuroplasticity is a fundamental brain process that underlies cognitive functioning and may give insight into the causes of cognitive dysfunction in TBI and schizophrenia. Neuroplasticity will be measured using electroencephalography (EEG) by placing small electrodes on the scalp that record the brain's electrical activity. Participants will listen to simple auditory tones and view simple visual patterns while their EEG is recorded. Additionally, participants will have measures of cognition and clinical interviews for diagnosis of a disorder as well as any current levels of symptoms.

DETAILED DESCRIPTION:
EEG recording: In this procedure, the participant's brain function will be recorded while listening to auditory tones or viewing simple visual stimuli. Participants will respond with a button press to specific tones or images. Participants will have all tasks clearly described to them and will practice each task prior to beginning the experiments. While performing these tasks, the brain's electrical activity (commonly referred to as "brain waves") will be recording using electroencephalography (EEG). Participant's will wear a cap that contains several electrodes (small, metal discs that are able to pick up electrical activity). A small amount of gel will be applied to the scalp underneath each electrode. These electrodes simply rest on the surface of the scalp and above and below the left eye. It takes approximately 15 minutes to place and prepare the electrodes. The entire recording session will last approximately 90 minutes (including setup). Before having EEG recorded it is important to wash the hair and scalp and not use conditioners or products in the hair as these may interfere with the electrical signal. The gel used is simply washed out of the hair with running water.

During the auditory task, participants will listen to a series of tones while watching a silent movie. Participants do not need to pay attention to the tones. During the visual task, participants will view a series of images on a computer screen that consist of a checkerboard pattern. Periodically, they will be asked to respond with a button press if one of the images is different than the others.

Interviews: There will be interviews conducted by trained staff that ask questions about participants' demographics (age, gender, education). A clinical interview will be given to all participants to determine if participants have either schizophrenia, a history of a traumatic brain injury, or have no psychiatric illness. All participants will be asked questions about how they are feeling. In addition, participants will answer questions about their family and friends and how they have been getting along with people in their lives.

Behavioral testing: Participants will have measures of cognition assessed using various computer-based tasks and pen-and-pencil questionnaires. These tests assess aspects of cognition including memory, attention, language, and motor skills. Participants will also be asked to view a series of pictures of faces and identify the emotion depicted on the face. Finally, participants will be asked to view a series of short videos consisting of a person telling a personal story. Participants will continuously rate how they think that person in the video is feeling (happy, sad, angry, etc.) while telling their story.

Additional Information: It may sometimes be necessary to contact a participant's physician to inquire about their medical history or diagnosis. Permission will be sought from participant's in order for contact to be made with their physician.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with a diagnosis of schizophrenia or a history of mild or moderate traumatic brain injury (TBI)
* Veterans without a psychiatric diagnosis and no history of TBI (healthy control participants) will also be recruited
* No other neurological or medical condition interfering with providing informed consent or valid assessment
* No current depression based on the Structured Clinical Interview for DSM-5 (SCID-I) or depressive symptoms rated moderate or higher

  * a rating of 13 or higher on the Hamilton Depression Rating Scale
* No DSM-V substance use disorder greater than mild severity in the past 3 months
* No form of cognitive remediation in the 6 months prior to testing
* An 8th grade reading level assessed with the Wide Range Achievement Test (WRAT)
* Normal or corrected-to-normal vision and hearing

Exclusion Criteria:

Exclusion criteria for all patient participants include:

* changes in medication dosage or type 3 months prior to testing
* hospitalization for psychiatric health in the 3 months prior to testing
* changes in housing status in the 6 months prior to testing

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wynn, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Green Lab — http://greenlab.dgsom.ucla.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | People With Schizophrenia | People With TBI | Healthy Controls
Started | 28 | 34 | 31
Completed | 26 | 23 | 26
Not Completed | 2 | 11 | 5
Not completed — Lost to Follow-up | 1 | 4 | 1
Not completed — Did not meet inclusion criteria | 1 | 6 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | People With Schizophrenia | People With TBI | Healthy Controls | Total
Number analyzed (Participants) | 26 | 23 | 26 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (9.8) | 42.9 (12.9) | 49.1 (12.9) | 48.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 1 | 7
  Male | 20 | 23 | 25 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 7 | 19
  Not Hispanic or Latino | 20 | 17 | 19 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 7 | 15 | 36
  White | 12 | 11 | 8 | 31
  More than one race | 0 | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 23 | 26 | 75

OUTCOME MEASURES:

1. Primary Outcome: Mismatch Negativity (MMN) Amplitudes in Microvolts
Description: Electroencephalography (EEG) measures the brain's activity while viewing simple visual stimuli or listening to simple auditory tones. MMN is measured while listening to a series of auditory tones, and is derived as the difference in responses to common stimuli minus rare stimuli (e.g., stimuli presented 90% of the time minus stimuli presented 10% of the time). A more negative value indicates stronger MMN, a more positive value indicates a stronger Repetition Positivity (RP) to the Standard stimuli, and a more negative value indicates a stronger Deviant Negativity (DN) to the Deviant stimuli. The investigators examined the deviant negativity, repetition positivity, and the MMN (which is defined as the difference between the standard-deviant), at three different standard tone repetition sequences (2, 6, or 36). In each case, the RP, DN, and MMN get stronger (i.e., larger amplitude) as the number of standard repetitions (2, 6, 36) increase.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | People With Schizophrenia | People With TBI | Healthy Controls
Number analyzed (Participants) | 25 | 22 | 25
microvolts
  MMN2 | -0.59 (2.38) | -1.19 (1.88) | -0.41 (1.89)
  MMN6 | -0.65 (2.01) | -1.87 (1.98) | -1.75 (2.11)
  MMN36 | -1.14 (1.92) | -3.13 (2.42) | -2.90 (2.86)
  Standard2 | 0.04 (1.53) | -0.46 (1.43) | -0.91 (1.27)
  Standard6 | -0.15 (1.39) | -0.40 (1.23) | 0.34 (1.15)
  Standard36 | 0.16 (1.02) | 0.08 (1.34) | 0.35 (1.44)
  Deviant2 | -0.54 (1.82) | -1.66 (1.36) | -1.32 (1.73)
  Deviant6 | -0.80 (1.44) | -2.26 (1.60) | -1.40 (2.00)
  Deviant36 | -0.98 (1.69) | -3.05 (1.90) | -2.55 (2.19)

2. Primary Outcome: Visual Long-Term Potentiation (LTP) Task
Description: This LTP task compares visual evoked potentials (VEPs) derived from the EEG before and after a period of extended visual stimulation (tetanization). We measured VEP amplitudes to two different checkerboard patterns before (pre-) and at three time points after (post-) a 10-minute prolonged tetanization checkerboard. VEPs were measured to tetanized (i.e., the same stimuli used in the 10-minute tetanization) or not tetanized (a different checkerboard pattern than the one used in tetanization) stimuli, prior to baseline (pre-), and at 5- (Post 1), 10- (Post 2), and 15- (Post 3) minutes after tetanization. This resulted in 4 VEP measurements for each tetanized and non-tetanized checkerboard. We focused on relative changes from baseline for evidence of plasticity and input specificity (i.e., tetanized vs. non-tetanized stimuli) at each of the 3 post-tetanization time points.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: microvolt
Arm/Group | People With Schizophrenia | People With TBI | Healthy Controls
Number analyzed (Participants) | 24 | 22 | 23
microvolt
  Pre-tetanization | 0.295 (1.758) | 0.201 (1.530) | 0.274 (1.554)
  Post-tetanization 1 | 1.215 (1.601) | 1.145 (1.217) | 1.149 (1.316)
  Post-tetanization 2 | 0.677 (1.489) | 0.360 (1.563) | 0.662 (1.319)
  Post-tetanization 3 | 0.475 (1.803) | 0.226 (1.722) | 0.540 (1.508)
  Pre-NonTetanized | 0.207 (0.664) | 0.155 (1.378) | 0.049 (1.203)
  Post-NonTetanized 1 | 0.557 (0.978) | 0.197 (1.217) | 0.508 (1.271)
  Post-NonTetanized 2 | 0.465 (0.951) | 0.364 (1.515) | 0.334 (1.408)
  Post-NonTetanized 3 | 0.325 (0.857) | 0.705 (1.303) | 0.142 (1.054)

3. Secondary Outcome: Neurocognition
Description: The MATRICS Consensus Cognitive Battery (MCCB) measures cognition in seven different domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition) and provides a SINGLE summary t-score (age and gender corrected) of overall cognitive functioning. The range of T-scores for a normal control population is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better overall cognitive functioning.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | People With Schizophrenia | People With TBI | Healthy Controls
Number analyzed (Participants) | 24 | 22 | 24
t-score | 35.13 (15.18) | 45.32 (11.34) | 46.29 (12.42)

4. Secondary Outcome: Empathic Accuracy
Description: Participants watch 9, short video clips of a person recounting a personal story. The participant must continuously rate how the person in the video is feeling while telling the story. The participant's ratings are then correlated with the ratings of the person who was in the video rating how they felt recounting their story. The average correlation for the 9 videos is the dependent variable, with higher positive correlations indicating higher empathic accuracy.
Time Frame: 1 Day
Population: We are unable to analyze the data due to an error in the scoring script that is not fixable.
Groups:
- People With TBI: People with mild to moderate diagnosis of TBI
- Healthy Control: Participants without schizophrenia or any psychotic disorder, and without a TBI
Arm/Group | People With Schizophrenia | People With TBI | Healthy Control
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Community Integration
Description: Community integration will be assessed by administering the Community Integration Questionnaire, which has 3 sub-scores (home, social, and activities). A higher score indicates better community integration.
Time Frame: 1 Day
Population: A higher score indicates better functioning. CIQ-home ranges from 0-10, CIQ-social ranges from 0-12, and CIQ-activities ranges from 0-17.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | People With Schizophrenia | People With TBI | Healthy Controls
Number analyzed (Participants) | 25 | 22 | 24
score on a scale
  CIQ-home | 5.88 (3.046) | 6.05 (2.870) | 6.67 (2.461)
  CIQ-social | 7.24 (2.332) | 8.45 (2.385) | 8.96 (2.116)
  CIQ-activities | 3.00 (1.581) | 4.36 (1.56) | 3.96 (1.574)

6. Secondary Outcome: Ekman Facial Affect Identification
Description: Participants view a series of 56 faces depicting one of seven different emotions (happy, sad, surprised, angry, afraid, disgusted, and neutral). The total number correctly identified faces is the outcome measure, with higher scores indicating better performance. Scores range from 0-56, with 56 indicating 100% accurate facial affect identification.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: score on a scale (total out of 56)
Arm/Group | People With Schizophrenia | People With TBI | Healthy Controls
Number analyzed (Participants) | 25 | 22 | 25
score on a scale (total out of 56) | 42.4 (7.1) | 46.4 (5.9) | 44.6 (5.7)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Does not differ. Total number of participants reflect those who met inclusion criteria and completed the study.
Arm/Group | People With Schizophrenia | People With TBI | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/23 | 0/26

LIMITATIONS AND CAVEATS:
Limitations mainly revolved around the study being interrupted and participant flow by the COVID-19 pandemic. However, the investigators largely met recruitment goals and successfully completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT03995368/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT03995368/ICF_000.pdf